CLINICAL TRIAL: NCT02790645
Title: Randomized Crossover Clinical Trial in Patients With Type 1 Diabetes Treated With Continuous Subcutaneous Insulin Infusion to Assess the Impact of Telemedicine vs. Conventional Medical Care. Integral Clinical Impact and Cost
Brief Title: Telemedicine Program in Type 1 Diabetes and CSII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Andaluz Health Service (Other Government); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CSII TELEMEDICINE PROGRAM
Record Dates: First submitted 2016-02-09; First posted 2016-06-06 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; Health technologies; Continuous subcutaneous insulin infusion; Telemedicine; Glycemic variability; Inflammatory markers,; Oxidative stress; Depression; Quality of life; Cost-effectiveness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1a. Control (Other): Treatment with CSII (Accu-Chek Spirit®) and follow-face doctor visits (conventional treatment -SMC-) (6 months).
  Interventions: Other: Group 1a. Control
- Group 2a. Telemedicine program (Other): CSII (Accu-Chek Spirit®) and medical monitoring via telematics application (Emminens Conecta® System, Roche Diagnostics SL) (TM) (6 months).
  Interventions: Other: Group 2a. Telemedicine program
- Group 1b. Telemedicine program (Other): After a washout period of 3 months and the crossing, Group 1 begins with medical monitoring via telematics application (Emminens Conecta® System, Roche Diagnostics SL) (TM) (6 months).
  Interventions: Other: Group 1b.Telemedicine program
- Group 2b. Control (Other): After a washout period of 3 months and the crossing, Group 2 begins with face doctor visits (conventional treatment -SMC-) (6 months).
  Interventions: Other: Group 2b. Control

INTERVENTIONS:
Other: Group 2a. Telemedicine program — CSII (Accu-Chek Spirit®) and medical monitoring via telematics application (Emminens Conecta® System, Roche Diagnostics SL) (TM) (6 months).
  Arms: Group 2a. Telemedicine program
Other: Group 1a. Control — Treatment with CSII (Accu-Chek Spirit®) and follow-face doctor visits (conventional treatment -SMC-) (6 months).
  Arms: Group 1a. Control
Other: Group 1b.Telemedicine program — After a washout period of 3 months and the crossing, Group 1 begins with medical monitoring via telematics application (Emminens Conecta® System, Roche Diagnostics SL) (TM) (6 months).
  Arms: Group 1b. Telemedicine program
Other: Group 2b. Control — After a washout period of 3 months and the crossing, Group 2 begins with face doctor visits (conventional treatment -SMC-) (6 months) .
  Arms: Group 2b. Control

SUMMARY:
Diabetes mellitus is a chronic disease of high socio-health relevance for their clinical and economic implications (risk of complications, disability ...) (healthcare costs). Strict glycemic control and intensive treatment and support have shown long-term patient with type 1 diabetes mellitus (DM1) improved health. The intensive insulin therapy involves the administration of insulin through 3 or more injections per day (MDI), or through a continuous subcutaneous insulin infusion (CSII). New technologies applied to the treatment of DM1, such as telemedicine, could bring benefits to patients. The available scientific evidence to date shows that telemedicine systems have beneficial or neutral effects on glycemic control, expressed in terms of HbA1c in patients with type 1 diabetes treated with MDI or CSII. They have also shown not to worsen the quality of life and reduce the costs associated with the care of these subjects. However, studies published to date are generally short follow-up, small sample size, and have not evaluated other biological parameters such as glycemic variability, inflammatory markers and markers of oxidative stress as well as a psychological assessment including depression, anxiety, Diabetes-related distress and fear of hypoglycemia. It has been designed a randomized crossover 18 months in order to study the effect of a telemedicine program in a group of subjects with DM1 in CSII on clinical variables of metabolic control variables, including parameters of glycemic variability, markers of inflammation and oxidative stress, psychological variables and quality of life, and associated costs.

DETAILED DESCRIPTION:
Randomized crossover clinical trial about the impact of a telemedicine program (Emminens Conecta® System, Roche Diagnostics SL) vs. the conventional medical follow-face of 18 months for the care of patients with DM1 intensive treatment with CSII (Accu-Chek Spirit®, Roche SL).

Two groups: one group with interactive clinical monitoring through a telemedicine platform (TM) and other conventional medical follow-up group (SMC) during 6 months. Being a crossover trial, both groups passing through both conditions (TM and SMC) during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes over 2 years of development with C plasma levels <0.5 ng / ml, and ISCI treated for> 6 months peptide.
* Age between 16 and 65 years (inclusive).
* HbA1c <10%.
* Absence of concomitant drug therapy that could affect blood glucose levels.
* Absence of chronic renal failure, abnormal liver function tests, thyroid disease active (except properly replaced hypothyroidism).
* Absence of acute decompensation Ketotic at baseline.

Exclusion Criteria:

* type 2 diabetes.
* type 1 diabetes treated with multiple daily insulin injections.
* Women pregnant or planning pregnancy.
* severe macrovascular or microvascular complications
* disabling psychological disorders.
* No collaboration (not signed informed consent).

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-09; Primary Completion 2016-04 (Actual); Study Completion 2016-09-19 (Actual)

PRIMARY OUTCOMES:
Assessment of clinical and metabolic parameters (glycosylated hemoglobin-HbA1c- and glycemic variability-SD-). | Baseline: Group 1 and 2
Assessment of clinical and metabolic parameters (glycosylated hemoglobin-HbA1c- and glycemic variability-SD-). | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)

SECONDARY OUTCOMES:
Assessment of inflammatory markers (hs-CRP). | Baseline: Group 1 and 2
Assessment of inflammatory markers (IL-6). | Baseline: Group 1 and 2
Assessment of inflammatory markers (TNF-α). | Baseline: Group 1 and 2
Assessment of inflammatory markers (MCP-1). | Baseline: Group 1 and 2
Assessment of inflammatory markers (hs-CRP). | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of inflammatory markers (IL-6). | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of inflammatory markers (TNF-α). | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of inflammatory markers (MCP-1). | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of redox markers (CAT). | Baseline: Group 1 and 2
Assessment of redox markers (TBARS). | Baseline: Group 1 and 2
Assessment of redox markers (oxidized LDL). | Baseline: Group 1 and 2
Assessment of redox markers (CAT). | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of redox markers (TBARS). | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of redox markers (oxidized LDL). | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of quality of life with the DQOL | Baseline: Group 1 and 2
Assessment of quality of life with the DQOL | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of depression with the BDI-II | Baseline: Group 1 and 2
Assessment of depression with the BDI-II | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of anxiety with the STAI | Baseline: Group 1 and 2
Assessment of anxiety with the STAI | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of distress related to diabetes with the DDS | Baseline: Group 1 and 2
Assessment of distress related to diabetes with the DDS | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of treatment satisfaction with the DTSQ | Baseline: Group 1 and 2
Assessment of treatment satisfaction with the DTSQ | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of fear of hypoglycemia with the FH-15 | Baseline: Group 1 and 2
Assessment of fear of hypoglycemia with the FH-15 | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of cost-effectiveness with a structured interview designed by our research group of direct and indirect costs. | Baseline: Group 1 and 2; 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)
Assessment of cost-effectiveness with a structured interview designed by our research group of direct and indirect costs. | 6 months: Control (Group1a+Group 2b) vs Telemedicine ( Group 2a+ Group1b)

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Ruiz de Adana, MD, PhD, Principal Investigator — Andaluz Health Service

REFERENCES:
- [Background] Jansa M, Vidal M, Viaplana J, Levy I, Conget I, Gomis R, Esmatjes E. Telecare in a structured therapeutic education programme addressed to patients with type 1 diabetes and poor metabolic control. Diabetes Res Clin Pract. 2006 Oct;74(1):26-32. doi: 10.1016/j.diabres.2006.03.005. Epub 2006 Apr 18. PMID 16621113
- [Background] Blanchet KD. Telehealth and diabetes monitoring. Telemed J E Health. 2008 Oct;14(8):744-6. doi: 10.1089/tmj.2008.8483. No abstract available. PMID 18954243